CLINICAL TRIAL: NCT07100574
Title: Bacteria in Dental Plaque and Atheroma Plaque
Status: Recruiting | Type: Observational
Sponsor: Istanbul Saglik Bilimleri University (Other)
Responsible Party: Principal Investigator, Ayşe Toraman, associate professor, Istanbul Saglik Bilimleri University
Other Study IDs: 1417
Record Dates: First submitted 2024-10-10; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Gingival Inflammation; Dental Plaque; Atheroma Plaque; Oral Bacteria
MeSH Terms: conditions — Gingivitis; Dental Plaque | interventions — Dental Plaque Index

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients diagnosed with endarterectomy
  Interventions: Other: atheroma plaque; Other: dental plaque

INTERVENTIONS:
Other: atheroma plaque — During the endarterectomy procedure, samples will be collected for study from some of the atheroma plaques routinely taken for pathology from patients.
Other: dental plaque — Subgingival plaque samples will be collected from patients before the endarterectomy procedure.

SUMMARY:
Periodontitis is considered a focus of infection where oral bacteria, bacterial by-products or inflammatory mediators can interact with other parts of the organism via the blood. Periodontal pathogen components such as DNA, RNA or specific antigens of P. gingivalis, Aggregatibacter actinomycetemcomitans (A. actinomycetemcomitans), Treponema denticola (T. denticola), Fusobacterium nucleatum (F. nucleatum) or Campylobacter rectus have been isolated from different tissues such as atheroma plaques, placenta, amniotic sac and respiratory tract. It has been reported that periodontitis may contribute to endothelial dysfunction leading to the formation of atherosclerosis.

DETAILED DESCRIPTION:
Periodontitis is considered a focus of infection where oral bacteria, bacterial by-products or inflammatory mediators can interact with other parts of the organism via the blood. Periodontal pathogen components such as DNA, RNA or specific antigens of P. gingivalis, Aggregatibacter actinomycetemcomitans (A. actinomycetemcomitans), Treponema denticola (T. denticola), Fusobacterium nucleatum (F. nucleatum) or Campylobacter rectus have been isolated from different tissues such as atheroma plaques, placenta, amniotic sac and respiratory tract. It has been reported that periodontitis may contribute to endothelial dysfunction leading to the formation of atherosclerosis.

Severe chronic generalized periodontitis may result in systemic inflammation and endothelial dysfunction. Periodontal bacteria produce endotoxins in the form of lipopolysaccharide (LPS). Circulating LPS causes an early systemic inflammatory response in the intima.

The aim of this study is to assess the relationship between bacteria in atheroma plaque, and dental plaque in patients grouped using the new periodontal classification. In addition, the relationship between demographic findings and bacterial count and frequency will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with endarterectomy
* Not receiving chemotherapy
* Not having received this treatment before

Exclusion Criteria:

* Having systemic infection
* Patients with severe heart disease

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Endearterectomy diagnosed, dentate and edentulous patients
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Number of bacteria | through study completion, an average of 2 months
  Subgingival plaque
Number of bacteria | through study completion, an average of 2 months
  atheroma plaque

CONTACTS AND LOCATIONS:
Locations (1):
- Health Sciences University, Hamidiye Faculty of Dentistry, Department of Periodontology, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No